CLINICAL TRIAL: NCT00139724
Title: A Phase III Randomized, Double-Blind, Double Dummy, Multi-Center Study To Compare The Efficacy, Safety And Tolerability Of Tolterodine Extended Release Capsule With Tolterodine Immediate Release Tablet In Subjects With Symptoms Of Overactive Bladder
Brief Title: Evaluate Efficacy and Safety Of Tolterodine Extended Release Capsule Compared With Tolterodine Immediate Release Tablet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6121112
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

INTERVENTIONS:
Drug: tolterodine extended release capsule

SUMMARY:
To evaluate efficacy of tolterodine extended release formulation compared with immediate release formulation in subjects with symptoms of overactive bladder

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of overactive bladder.

Exclusion Criteria:

* Subjects with significant stress incontinence as determined by the investigator.
* Subjects with recurrent urinary tract infections defined as treated for UTI; 5 times in the last year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2005-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of tolterodine extended release formulation compared with immediate release formulation after 8 weeks of treatment in subjects with symptoms of overactive bladder

SECONDARY OUTCOMES:
To evaluate the safety of tolterodine extended release formulation compared with immediate release formulation after 8 weeks of treatment in subjects with symptoms of overactive bladder.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- China (5):
  - Pfizer Investigational Site, Beijing, Beijing Municipality
  - Pfizer Investigational Site, Huangzhou, Zhejiang
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Chongqing
  - Pfizer Investigational Site, Shanghai

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6121112&StudyName=Evaluate+Efficacy+and+Safety+Of+Tolterodine+Extended+Release+Capsule+Compared+With+Tolterodine+Immediate+Release+Tablet+